CLINICAL TRIAL: NCT04395144
Title: Randomized-controlled Trial of HFNC Alone vs HFNC and Awake Self-proning for Treatment of Severe COVID-19
Brief Title: COVid-19: Awake Proning and High-flow Nasal Cannula in respiratorY DistrEss
Acronym: COVAYDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital de Verdun (Other)
Responsible Party: Principal Investigator, Ivan Pavlov, Emergency physician, Hôpital de Verdun
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-01
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Coronavirus Infection; COVID; Severe Acute Respiratory Syndrome; Respiratory Failure; Respiratory Insufficiency; Respiratory Distress Syndrome; ARDS; Lung Diseases
Keywords: SARS-CoV-2; SARS-CoV-2 infection; COVID-19; HFNC; HFNO; Proning; Prone position; High-flow nasal cannula; High-flow nasal oxygenation; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Coronavirus Infections; Severe Acute Respiratory Syndrome; Respiratory Insufficiency; Respiratory Distress Syndrome; Lung Diseases; COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Awake prone positioning (Experimental): Prone positioning of patients on nasal high-flow oxygen therapy
  Interventions: Procedure: Awake Prone Positioning
- Standard care (Active Comparator): Standard decubitus positioning of patients on nasal high-flow oxygen therapy
  Interventions: Procedure: Standard care

INTERVENTIONS:
Procedure: Awake Prone Positioning — Patients will receive instruction to remain in prone position as long and as often as possible, up to 16h/24h
  Arms: Awake prone positioning
Procedure: Standard care — Patients will not receive any special instructions with regards to proning.
  Arms: Standard care

SUMMARY:
Prone positioning is an established intervention in mechanically ventilated acute respiratory distress syndrome (ARDS) patients, with demonstrated reductions in mortality.

Preliminary data suggest that awake proning in patients with COVID-19 treated with high-flow nasal oxygenation (HFNO) improves gas exchanges, and might be associated with a reduced need of mechanical ventilation, and reduced mortality. Further investigation in a formal randomized-controlled trial is need.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19, either confirmed by SARS-CoV-2 assay, or clinically suspected, with results of the assay pending;
* Lung infiltrates documented on chest X-ray or chest CT-scan;
* Significant respiratory distress that requires treatment with HFNO.

Exclusion Criteria:

* Unable to consent;
* Unable to prone;
* Indication for immediate endotracheal intubation and mechanical ventilation;
* Contraindication to prone positioning (severe obesity, abdominal wound, pregnancy, unstable pelvic/spinal lesions, vomiting, etc.);
* Comfort care or imminent expectation of death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Rate of Therapeutic failure, defined as a combined outcome of rate of intubation or death | Up to 28 days after randomization

SECONDARY OUTCOMES:
Intubation rate | Up to 28 days after randomization
Mortality | Up to 28 days after randomization
Days spent on mechanical ventilation | Until discharge, up to 24 weeks after randomization
Days spent in the ICU | Until discharge, up to 24 weeks after randomization
Hospital stay (in days) | From admission to discharge, up to 24 weeks after randomization

OTHER OUTCOMES:
Time in prone position | Up to 28 days post randomization
  Total time spent in prone position, as recorded by nursing or respiratory therapists
Oxygenation (SpO2/FiO2 ratio) | Until HFNC weaning, or up to 14 days after randomization, whichever is first
  Daily evolution of oxygenation

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Pavlov, MD, Principal Investigator — Hôpital de Verdun
Locations (5):
- Canada (5):
  - Hôtel-Dieu de Gaspé, Gaspé, Quebec
  - Hôpital de la Cité-de-la-Santé, Laval, Quebec
  - Montreal General Hospital, McGill University Healthcare Center, Montreal, Quebec
  - Royal Victoria Hospital, McGill University Healthcare Center, Montreal, Quebec
  - Hôpital de Verdun, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ehrmann S, Li J, Ibarra-Estrada M, Perez Y, Pavlov I, McNicholas B, Roca O, Mirza S, Vines D, Garcia-Salcido R, Aguirre-Avalos G, Trump MW, Nay MA, Dellamonica J, Nseir S, Mogri I, Cosgrave D, Jayaraman D, Masclans JR, Laffey JG, Tavernier E; Awake Prone Positioning Meta-Trial Group. Awake prone positioning for COVID-19 acute hypoxaemic respiratory failure: a randomised, controlled, multinational, open-label meta-trial. Lancet Respir Med. 2021 Dec;9(12):1387-1395. doi: 10.1016/S2213-2600(21)00356-8. Epub 2021 Aug 20. PMID 34425070
- [Derived] Tavernier E, McNicholas B, Pavlov I, Roca O, Perez Y, Laffey J, Mirza S, Cosgrave D, Vines D, Frat JP, Ehrmann S, Li J. Awake prone positioning of hypoxaemic patients with COVID-19: protocol for a randomised controlled open-label superiority meta-trial. BMJ Open. 2020 Nov 11;10(11):e041520. doi: 10.1136/bmjopen-2020-041520. PMID 33177145